CLINICAL TRIAL: NCT01654029
Title: Patient Centred Communication Intervention
Acronym: PCCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCCI 93790
Record Dates: First submitted 2012-07-20; First posted 2012-07-31 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Aphasia; Stroke
Keywords: Stroke; Communication impairments; Nurse-patient communication; Patient-centred care
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group receiving usual care (No Intervention): Usual care consists of speech language therapy for some patients. Most care is focused on swallowing assessments.
- PCCI Intervention (Experimental): The Patient-Centred Communication Intervention consists of 1) development of a communication care plan; 2)a workshop for staff focused on communication and behavioural management strategies,: and 3) implementing a staff support system.
  Interventions: Behavioral: Patient-Centred Communication Intervention

INTERVENTIONS:
Behavioral: Patient-Centred Communication Intervention — The intervention consists of three parts: 1) development of individualized communication care plans; 2) staff attendance at a workshop focused on communication and behavioral management strategies; and 3) implementation of a staff support system.
  Arms: PCCI Intervention

SUMMARY:
The most frequent consequence of a stroke is a communication impairment. When patients cannot articulate their needs, frustration and agitation are frequent responses, often resulting in poor optimization of post-stroke function. Staff's lack of knowledge of communication strategies exacerbates the problem. A key component of patient-centred care is the ability of staff to communicate in such a way that allows them to understand the patient's needs. Members of our team developed the patient-centred communication intervention (PCCI) targeting registered and unregulated staff caring for complex continuing care (CCC) patients with communication impairments post stroke. The purpose of the study is to examine if the PCCI results in improved patients' quality of life and in improved staff attitudes and skills in caring for patients with communication impairments.

ELIGIBILITY:
Patients:

Inclusion Criteria

* diagnosis of stroke related to cerebral infarct
* presence of a communication impairment
* ability to speak and understand English before the stroke
* ability to consent

Exclusion Criteria:

* global aphasia or severe Wernicke's aphasia

Staff:

Inclusion Criteria

* directly involved in providing care
* employed full or part-time
* ability to consent
* ability to speak and write English
* work with patients who have communication impairments

Exclusion Criteria

* unwilling to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Stroke and Aphasia Quality of Life (SAQOL) | Change in SAQOL from baseline to 1 month and from baseline to 3 months
  The SAQOL is a 39-item tool designed to measure health-related quality of life in patients post-stroke with aphasia.

SECONDARY OUTCOMES:
Communication-Impairment Questionnaire (CIQ) | Change in CIQ from baseline to 1 month and from baseline to 3 months
  The Communication Impairment Questionnaire is an 8-item self-report scale. It is used to measure the attitudes of nurses toward patients with communication impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine S McGilton, RN, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute, E.W. Bickle Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] McGilton KS, Sorin-Peters R, Sidani S, Boscart V, Fox M, Rochon E. Patient-centred communication intervention study to evaluate nurse-patient interactions in complex continuing care. BMC Geriatr. 2012 Oct 11;12:61. doi: 10.1186/1471-2318-12-61. PMID 23050517